CLINICAL TRIAL: NCT04914481
Title: AnaTomic Stenosis Severity Derived From Computed Tomography as a Prognostic Marker in Patients With Low-flow Low-gradient Aortic Stenosis Undergoing Transcatheter Aortic Valve Implantation
Brief Title: Anatomic Stenosis Severity as a Prognostic Marker in Patients With Low-Flow Low-Gradient Aortic Stenosis Undergoing TAVI
Acronym: ATLAS TAVI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Sponsor
Other Study IDs: ATLAS TAVI
Record Dates: First submitted 2021-06-02; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Low-Flow, Low-Gradient Aortic Stenosis
Keywords: Aortic Stenosis; Low-Flow, Low-Gradient; TAVI
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Classical Low-Flow, Low-Gradient Aortic Stenosis: Classical Low-Flow, Low-Gradient Aortic Stenosis is defined as valve area <1 cm2, mean gradient <40 mmHg, ejection fraction <50% and stroke volume index (SVi) ≤35 mL/m2 by resting transthoracic echocardiography. Dobutamine stress echocardiography is not mandatory for the definition of classical LFLG AS. All patients in this subgroup underwent TAVI and have available data on aortic valve calcification.
- Paradoxical Low-Flow, Low-Gradient Aortic Stenosis: Paradoxical Low-Flow, Low-Gradient Aortic Stenosis is defined as valve area <1 cm2, mean gradient <40 mmHg, ejection fraction ≥50% and SVi ≤35 mL/m2 by resting transthoracic echocardiography. All patients in this subgroup underwent TAVI and have available data on aortic valve calcification.
- High-Gradient Aortic Stenosis (Control group): High-Gradient Aortic Stenosis is defined as valve area <1 cm2 and mean gradient >40 mmHg by resting transthoracic echocardiography. All patients in this subgroup underwent TAVI. Data on aortic valve calcification is not mandatory for this control group.
- Conservative treatment (Control group): The subgroup includes all patients with (severe or non-severe) aortic stenosis, who underwent conservative treatment. Data on aortic valve calcification is not mandatory for this control group.

SUMMARY:
The ATLAS TAVI Registry is a retrospective, investigator-initiated, multicenter registry including patients, who underwent Transcatheter Aortic Valve Implantation (TAVI) for classical or paradoxical low-flow, low-gradient aortic stenosis (LFLG AS) with available non-contrast MSCT data on aortic valve calcification (AVC). The main objective of this study is the assessment of outcome after TAVI according to AVC density severity in patients with LFLG AS.

DETAILED DESCRIPTION:
Aortic valve calcification (AVC) as assessed by MSCT is highly correlated with aortic stenosis (AS) severity and, thus, has become an important tool for diagnosing severe AS, especially in patients with low-flow low-gradient aortic stenosis (LFLG AS). Moreover, in medically treated AS patients AVC is directly associated with poor prognosis. In contrast, the prognostic benefit of eliminating AS by Transcatheter Aortic Valve Implantation (TAVI) in patients with LFLG AS seems to be larger in patients with high AVC density (AVCd) compared to those with low AVCd, at least in "classical" (low EF) LFLG AS. Hence, we hypothesize that AVCd might be a valuable marker for treatment response among TAVI patients with LFLG AS, who are known to suffer from poor outcome even after elimination of AS.

The multicentric ATLAS TAVI Registry of LFLG AS patients, who underwent TAVI, assesses the impact of AVCd on outcome in these patients.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* patient gave written informed consent for data acquisition and transfer
* for LFLG AS: -- available non-contrast MSCT data on aortic valve calcification (AVC, Agatston Units)

Exclusion Criteria:

- LFLG AS without non-contrast MSCT data on AVC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective, investigator-initiated, multicenter registry including patients, who underwent TAVI for classical or paradoxical LFLG AS with available non-contrast MSCT data on AVC. Furthermore, data will be gathered for the control groups of patients with high-gradient AS, who underwent TAVI, and heart failure patients with concomitant AS, who underwent medical treatment. MSCT data will not be mandatory for control groups.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 12 months

SECONDARY OUTCOMES:
Cardiovascular Mortality | 12 months
  Incidence of cardiovascular death, defined as death attributable to myocardial ischemia and infarction, heart failure, cardiac arrest because of other or unknown cause, or cerebrovascular accident.
Rehospitalizations for congestive heart failure | 12 months
  Incidence of new-onset or worsening signs and symptoms of heart failure that required urgent therapy and resulted in hospitalization, e.g. as assessed by patient interviews or hospital records.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Annick Clavel, PhD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Canada; Niklas Schofer, MD, Principal Investigator — University Heart and Vascular Center Hamburg, Hamburg, Germany; Sebastian Ludwig, MD, Principal Investigator — University Heart and Vascular Center Hamburg, Hamburg, Germany
Locations (11):
- Canada (2):
  - Montreal Heart Institute, Montreal
  - Institut universitaire de cardiologie et de pneumologie de Québec, Université Laval, Québec
- Odense University Hospital, Odense, Denmark
- France (2):
  - CHU de Lille, Lille
  - Hôpital Bichat - Claude-Bernard, Paris
- Germany (3):
  - Kerckhoff-Klinik, Bad Nauheim
  - University Heart and Vascular Center Hamburg, Hamburg
  - Heart Center Leipzig, Leipzig
- Rabin Medical Center, Petah Tikva, Israel
- Erasmus University Medical Centre, Rotterdam, Netherlands
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cueff C, Serfaty JM, Cimadevilla C, Laissy JP, Himbert D, Tubach F, Duval X, Iung B, Enriquez-Sarano M, Vahanian A, Messika-Zeitoun D. Measurement of aortic valve calcification using multislice computed tomography: correlation with haemodynamic severity of aortic stenosis and clinical implication for patients with low ejection fraction. Heart. 2011 May;97(9):721-6. doi: 10.1136/hrt.2010.198853. Epub 2010 Aug 18. PMID 20720250
- [Background] Clavel MA, Messika-Zeitoun D, Pibarot P, Aggarwal SR, Malouf J, Araoz PA, Michelena HI, Cueff C, Larose E, Capoulade R, Vahanian A, Enriquez-Sarano M. The complex nature of discordant severe calcified aortic valve disease grading: new insights from combined Doppler echocardiographic and computed tomographic study. J Am Coll Cardiol. 2013 Dec 17;62(24):2329-38. doi: 10.1016/j.jacc.2013.08.1621. Epub 2013 Sep 24. PMID 24076528
- [Background] Clavel MA, Pibarot P, Messika-Zeitoun D, Capoulade R, Malouf J, Aggarval S, Araoz PA, Michelena HI, Cueff C, Larose E, Miller JD, Vahanian A, Enriquez-Sarano M. Impact of aortic valve calcification, as measured by MDCT, on survival in patients with aortic stenosis: results of an international registry study. J Am Coll Cardiol. 2014 Sep 23;64(12):1202-13. doi: 10.1016/j.jacc.2014.05.066. PMID 25236511
- [Background] Ludwig S, Gossling A, Waldschmidt L, Linder M, Bhadra OD, Voigtlander L, Schafer A, Deuschl F, Schirmer J, Reichenspurner H, Blankenberg S, Schafer U, Westermann D, Seiffert M, Conradi L, Schofer N. TAVR for low-flow, low-gradient aortic stenosis: Prognostic impact of aortic valve calcification. Am Heart J. 2020 Jul;225:138-148. doi: 10.1016/j.ahj.2020.03.013. Epub 2020 Apr 8. PMID 32502877
- [Background] Baumgartner H, Falk V, Bax JJ, De Bonis M, Hamm C, Holm PJ, Iung B, Lancellotti P, Lansac E, Rodriguez Munoz D, Rosenhek R, Sjogren J, Tornos Mas P, Vahanian A, Walther T, Wendler O, Windecker S, Zamorano JL; ESC Scientific Document Group. 2017 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2017 Sep 21;38(36):2739-2791. doi: 10.1093/eurheartj/ehx391. No abstract available. PMID 28886619
- [Derived] Ludwig S, Schofer N, Abdel-Wahab M, Urena M, Jean G, Renker M, Hamm CW, Thiele H, Iung B, Ooms JF, Wiessman M, Mogensen NSB, Longere B, Perrin N, Ben Ali W, Coisne A, Dahl JS, Van Mieghem NM, Kornowski R, Kim WK, Clavel MA. Transcatheter Aortic Valve Replacement in Patients With Reduced Ejection Fraction and Nonsevere Aortic Stenosis. Circ Cardiovasc Interv. 2023 May;16(5):e012768. doi: 10.1161/CIRCINTERVENTIONS.122.012768. Epub 2023 May 16. PMID 37192310